CLINICAL TRIAL: NCT01553409
Title: Prospective Observational Study on the Effects of Blood Donation on Blood Pressure, Iron Metabolism and Oxidative Stress
Brief Title: Effect of Blood Donation on Blood Pressure, Iron Metabolism, Oxidative Stress
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Chair of clinical naturopathic medicine, Charite University, Berlin, Germany
Other Study IDs: 89834103
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
Keywords: Hypertension; Ferritin; Phlebotomy; Blood donation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — regular blood donation is done and from blood, that is taken for blood tests by the blood donation center any there are made blood tests of lipid metabolism, iron metabolism and antioxidative stress
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators want to investigate the effects of blood donation to blood pressure, to iron metabolism and oxidative stress.

There are results of other studies that show, that there is a positive effect of blood donation to high blood pressure, iron metabolism and oxidative stress.

DETAILED DESCRIPTION:
The regular application flow of blood donation at that blood bank of Charité is not disturbed. There are only some more questions and measurement of blood pressure, iron metabolism, fat metabolism and oxidative stress.

No extra puncture of the vein is necessary.

ELIGIBILITY:
Inclusion Criteria:

* first time donating blood or after a break of 12 months to last blood donation
* voluntary attending blood donation and study
* fulfilling the criteria of the blood donation center

Exclusion Criteria:

* criteria of the blood donation center (e. g. low haemoglobin, fever, acute infection, having spent in tropical countries for the last months,general bad health condition,...)
* missing informed consent to the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: female and male from 18 years to 65 years, who are able and want to donate blood for the first time or after one year break to the last blood donation
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
blood pressure | 3 months
  seated blood pressure will be measured baseline and after 3 months by trained professionals

SECONDARY OUTCOMES:
blood pressure | 12 months
  seated blood pressure will be measured baseline and after 12 months by trained professionals

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charite University; Abdulgabar Salama, Prof. Dr., Principal Investigator — Charite University
Locations (1):
- Charité Universitätsmedizin Berlin Blutspende Campus Mitte, Berlin, Germany